CLINICAL TRIAL: NCT07128446
Title: Development and Feasibility Evaluation of Canadian Occupational Performance Measure-Based Goal Setting Strategies for Pediatric Intensive Care Unit Patients: A Multi-Phase Mixed-Methods Study
Brief Title: COPM-Based Goal Setting Strategies in the PICU
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Jeong Yi Kwon, Professor, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-08-032
Record Dates: First submitted 2025-08-13; First posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Critical Illness; Pediatric Intensive Care Unit
MeSH Terms: conditions — Critical Illness | interventions — Occupational Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Standard physical and occupational therapy (Experimental): Participants will receive standard physiacal and occupational therapy as routinely provided in the PICU. The therapy may include activities of daily living training, positioning, range of motion exercises, and caregiver education, according to each patient's condition. No experimental intervention is introduced; the study focuses on evaluating patient-centered outcomes using the Canadian Occupational Performance Measure.
  Interventions: Other: Standard physical and occupational therapy

INTERVENTIONS:
Other: Standard physical and occupational therapy — Participants admitted to the Pediatric Intensive Care Unit (PICU) will receive standard occupational therapy as part of routine clinical care. Interventions will be tailored to each patient's medical status and functional needs and may include activities of daily living (ADL) training, positioning, range of motion exercises, sensory stimulation, and caregiver education. No additional experimental treatment will be introduced for study purposes. The primary focus of the study is to evaluate patient-centered outcomes using the Canadian Occupational Performance Measure (COPM), without altering the standard therapeutic approach.

SUMMARY:
COPM-Based Goal Setting Strategies in the PICU

ELIGIBILITY:
Inclusion Criteria:

Phase 1-2 (Delphi Survey - Experts)

* Physicians specializing in pediatrics or physical medicine and rehabilitation, occupational therapists, physical therapists, and nursing staff
* Minimum of 2 years of direct clinical experience in a Pediatric Intensive Care Unit (PICU)

Phase 3 (Pilot Testing - Caregivers & PICU Clinicians)

Caregivers:

* Legal guardian of a child aged 1-18 years admitted to PICU
* ≥24 hours post-admission

PICU clinicians:

- Treating occupational or physical therapist involved in the child's care during PICU admission

Exclusion Criteria:

Phase 1-2 (Delphi Survey - Experts)

* Rehabilitation professionals without prior PICU clinical experience
* Inability to read or respond to Korean-language surveys

Phase 3 (Pilot Testing - Caregivers & PICU Clinicians)

* Caregivers experiencing severe emotional distress, or deemed inappropriate for participation by the treating clinician
* Non-Korean-speaking caregivers
* Refusal or withdrawal of informed consent at any stage

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 5 (Estimated)
Dates: Start 2025-09-20 (Estimated); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Consensus Level for COPM Implementation Criteria in the PICU (Delphi Survey) | From initial Delphi invitation to completion of second round (estimated 2-3 weeks).
  Level of expert consensus on specific clinical and procedural criteria for implementing COPM-based goal-setting in PICU, measured via a two-round online Delphi survey. Consensus is defined as ≥70% agreement (≥6/10 on a Likert scale) and mean score ≥7 for Likert items, or ≥50% selection for categorical items.

SECONDARY OUTCOMES:
Client-Centredness of Goal Setting (C-COGS) | Immediately after pilot intervention completion.
  C-COGS questionnaire will assess the extent to which client-centred principles are reflected in goal-setting for PICU caregivers. The tool includes 13 items across two subscales: Participation (9 items, max 45 points) and Goal Subscale (up to 24 items). Total scores range from 0-50, with higher scores indicating greater client-centredness.
Caregiver Perceived Acceptability and Feasibility of COPM-Based Goal Setting in PICU | Immediately after pilot intervention completion.
  Structured survey developed for this study, based on items from MPOC-20, to assess caregiver perceptions of acceptability, feasibility, and perceived clinical relevance of the COPM-based goal-setting strategy. The survey includes 9 items (7 quantitative on 5-point Likert scale, 2 open-ended for qualitative analysis). Higher scores indicate greater perceived acceptability and feasibility.

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared. The dataset includes sensitive clinical information from PICU patients and their caregivers. Due to concerns about patient privacy, potential re-identification risk, and institutional review boardrestrictions, IPD will be used solely for the purposes defined in the approved protocol and will not be made available for external access.

REFERENCES:
- [Result] Hwang Y, Kwon JY, Cho J, Choi J. Individualized Goal Setting for Pediatric Intensive Care Unit-Based Rehabilitation Using the Canadian Occupational Performance Measure. Children (Basel). 2023 May 31;10(6):985. doi: 10.3390/children10060985. PMID 37371217